CLINICAL TRIAL: NCT02745119
Title: A Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of Lampalizumab in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration Who Have Completed a Roche-Sponsored Study
Brief Title: Long-Term Safety of Lampalizumab Intravitreal (ITV) Injections in Participants With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (OMASPECT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX30191; 2016-000423-13 (EudraCT Number)
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-01

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — lampalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lampalizumab Every 4 Weeks (Experimental): Participants who received either lampalizumab or sham comparator every 4 weeks in one of the parent studies and completed the Week 96 visit will receive open-label lampalizumab as 10 milligrams (mg) via ITV injection, administered every 4 weeks.
  Interventions: Drug: Lampalizumab
- Lampalizumab Every 6 Weeks (Experimental): Participants who received either lampalizumab or sham comparator every 6 weeks in one of the parent studies and completed the Week 96 visit will receive open-label lampalizumab as 10 mg via ITV injection, administered every 6 weeks.
  Interventions: Drug: Lampalizumab

INTERVENTIONS:
Drug: Lampalizumab — Lampalizumab 10 mg will be administered every 4 or 6 weeks according to the frequency given during participation in the parent study.

SUMMARY:
This multicenter open-label extension study is designed to evaluate the safety and tolerability of lampalizumab intravitreal injections in participants with GA secondary to age-related macular degeneration (AMD) who completed 96 weeks of treatment in Studies GX29176 (NCT02247479) or GX29185 (NCT02247531). The extension will enroll participants from the parent studies who received investigational lampalizumab, as well as lampalizumab-naive participants exposed to sham comparator. All participants will receive open-label lampalizumab in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in Studies GX29176 (NCT02247479) or GX29185 (NCT02247531) with completion of treatment and the Week 96 visit
* Agreement to remain abstinent or use a reliable form of contraception among all men and among women of child-bearing potential

Exclusion Criteria:

* Concurrent ocular conditions that contraindicate use of lampalizumab or might affect interpretation of study results or that might increase the risk of treatment complications
* Concurrent disease, metabolic dysfunction, or physical or laboratory finding that contraindicates use of lampalizumab or might affect interpretation of study results or that might increase the risk of treatment complications
* Increased risk of infection
* Pregnancy or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 994 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (208):
- United States (122):
  - Uni of Alabama At Birmingham Clinical Research Unit, Birmingham, Alabama
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Retina Centers P.C., Tucson, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Consultants of Orange County, Fullerton, California
  - UCSD Shiley Eye Center, La Jolla, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - N CA Retina Vitreous Assoc, Mountain View, California
  - East Bay Retina Consultants, Oakland, California
  - Southern CA Desert Retina Cons, Palm Desert, California
  - Byers Eye Insitute at Stanford, Palo Alto, California
  - Retina Consultants, San Diego, Poway, California
  - University of California, Davis, Eye Center, Sacramento, California
  - Retinal Consultants Med Group, Sacramento, California
  - W Coast Retina Med Group Inc, San Francisco, California
  - UCSF Comprehensive Cancer Ctr; Ophthalmology, San Francisco, California
  - Orange County Retina Med Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - University of Colorado, Aurora, Colorado
  - Retina Consultants of Southern, Colorado Springs, Colorado
  - Colorado Retina Associates, PC, Golden, Colorado
  - Retina Group of New England, New London, Connecticut
  - Florida Eye Microsurgical Inst, Boynton Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Retina Health Center, Fort Myers, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Bascom Palmer Eye Institute, Naples, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Midwest Eye Institute Northside, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, Shawnee Mission, Kansas
  - Vitreo Retinal Consultants, Wichita, Kansas
  - Lahey Clinic Med Ctr, Lexington, Kentucky
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Wilmer Eye Institute, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Retina Specialists, Towson, Maryland
  - Tufts Medical Center Research, Boston, Massachusetts
  - Mass Eye and Ear Infirmary, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Kresge Eye Institute, Detroit, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Specialty Eye Institute, Jackson, Michigan
  - Assoc Retinal Consultants PC, Royal Oak, Michigan
  - Retina Consultants of Michigan, Southfield, Michigan
  - Vitreoretinal Surgery, Edina, Minnesota
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Retina Consultants of Nevada, Las Vegas, Nevada
  - Sierra Eye Associates, Reno, Nevada
  - Retina Center of New Jersey, Bloomfield, New Jersey
  - Mid Atlantic Retina - Wills Eye Hospital, Cherry Hill, New Jersey
  - New Jersey Retina Research Foundation, Edison, New Jersey
  - Delaware Valley Retina Assoc, Lawrenceville, New Jersey
  - Retinal & Ophthalmic Cons PC, Northfield, New Jersey
  - Retina Associates of NJ, Teaneck, New Jersey
  - Lions Eye Institute, Albany, New York
  - Long Is. Vitreoretinal Consult, Hauppauge, New York
  - Opthalmic Consultants of LI, Lynbrook, New York
  - New York Eye & Ear Infirmary, New York, New York
  - Vitreous-Retina-Macula, New York, New York
  - Retina Assoc of Western NY, Rochester, New York
  - Retina Vit Surgeons/Central NY, Syracuse, New York
  - West Carolina Retinal AssocPA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Duke University Eye Center; Vitreoretinal, Durham, North Carolina
  - Wake Forest Baptist Health Eye Centre, Winston-Salem, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Assoc of Cleveland Inc, Cleveland, Ohio
  - Cleveland Clinic Foundation; Cole Eye Institute, Cleveland, Ohio
  - OSU Eye Physicians & Surgeons, Columbus, Ohio
  - Retina & Vitreous Center of Southern Oregon, Ashland, Oregon
  - Retina Northwest, Portland, Oregon
  - Oregon HSU; Casey Eye Institute, Portland, Oregon
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Associates in Ophthalmology, West Mifflin, Pennsylvania
  - Palmetto Retina Center, Florence, South Carolina
  - Charleston Neuroscience Inst, Ladson, South Carolina
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Charles Retina Institution, Germantown, Tennessee
  - Tennessee Retina PC., Nashville, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Valley Retina Institute P.A., McAllen, Texas
  - Scott and White Hospital, Temple, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Univ of Virginia Ophthalmology, Charlottesville, Virginia
  - Eye Surgeons of Richmond Inc. dba Virginia Eye Institute, Richmond, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Virginia Retina Center, Warrenton, Virginia
  - Vitreoretinal Associates of Washington, Bellevue, Washington
  - Retina Center Northwest, Silverdale, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - West Virginia University Eye Institute, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Australia (6):
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Marsden Eye Research Centre, Parramatta, New South Wales
  - Save Sight Institute, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - Vision Eye Institute Eastern, Box Hill, Victoria
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
- Austria (2):
  - Kepler Universitätskliniken GmbH - Med Campus III; Abt. für Augenheilkunde, Linz
  - Medizinische Universität Wien; Universitätsklinik für Augenheilkunde und Optometrie, Vienna
- Belgium (2):
  - CHU Brugmann (Victor Horta), Brussels
  - UZ Leuven Sint Rafael, Leuven
- Institut De L'Oeil Des Laurentides, Boisbriand, Quebec, Canada
- Denmark (2):
  - Glostrup Hospital, Øjenafdelingen, Forskningsafsnit Ø37, Glostrup Municipality
  - Sjællands Universitetshospital, Roskilde; Øjenafdelingen, Roskilde
- France (7):
  - Hopital Pellegrin; Ophtalmologie, Bordeaux
  - Chi De Creteil; Ophtalmologie, Créteil
  - Hôpital de La Croix Rousse, Lyon
  - Centre Monticelli Paradis d Ophtalmologie, Marseille
  - CHU Nantes - Hôtel Dieu; Ophthalmology, Nantes
  - Centre Odeon; Exploration Ophtalmologique, Paris
  - CHNO des Quinze Vingts; Ophtalmologie, Paris
- Germany (13):
  - Universitäts-Augenklinik Bonn, Bonn
  - Universitätsklinikum Köln; Augenklinik, Cologne
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Klinik für Augenheilkunde, Hanover
  - Universitätsklinik Heidelberg; Augenklinik, Heidelberg
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH; Augenklinik, Ludwigshafen
  - Universitätskliniikum Schleswig-Holstein, Campus Lübeck, Klinik für Augenheilkunde, Lübeck
  - LMU Klinikum der Universität, Augenklinik, München
  - Klinikum rechts der Isar der TU München; Augenklinik, München
  - Augenabteilung am St. Franziskus-Hospital, Münster
  - Universitätsklinikum Münster; Augenheilkunde, Münster
  - Universitätsklinikum Regensburg, Klinik & Poliklinik für Augenheilkunde, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (5):
  - Semmelweis Egyetem AOK, Szemeszeti Klinika, Budapest
  - Budapest Retina Associates Kft., Budapest
  - Peterfy Sandor utcai Korhaz-Rendelointezet es Baleseti Kozpont, Szemeszet KR, Budapest
  - Debreceni Egyetem Klinikai Kozpont; Szemeszeti Klinika, Debrecem
  - Ganglion Medial Center, Pécs
- Italy (6):
  - Fondazione Ptv Policlinico Tor Vergata Di Roma;U.O.S.D. Patologie Renitiche, Rome, Lazio
  - UNIVERSITA' DEGLI STUDI DI GENOVA - Di.N.O.G.;CLINICA OCULISTICA, Genoa, Liguria
  - Irccs Ospedale San Raffaele;U.O. Oculistica, Milan, Lombardy
  - ASST FATEBENEFRATELLI SACCO; Oculistica (Sacco), Milan, Lombardy
  - A.S.L. to1 Presidio Ospedaliero Sperino Oftalmico, Turin, Piedmont
  - A.O. Universitaria S. Maria Della Misericordia Di Udine; Clinica Oculistica, Udine, Veneto
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- TG Laser Oftalmica, Lima, Peru
- Poland (7):
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Szpital Specjalistyczny nr 1; Oddzial Okulistyki, Bytom
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddział Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
  - Klinika Okulistyczna Jasne Błonia, Lodz
  - Uniwersytecki Szpital Kliniczny; Klinika Okulistyki, Wroclaw
- Portugal (3):
  - AIBILI - Association for Innovation and Biomedical Research on Light, Coimbra
  - Espaco Medico Coimbra, Coimbra
  - Hospital de Santa Maria; Servico de Oftalmologia, Lisbon
- Slovakia (4):
  - Nemocnica sv. Michala, a.s., Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica sv. Cyrila a Metoda Ocna klinika SZU a UNB, Bratislava
  - Fakultna nemocnica Trencin Ocna klinika, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina; Ocne oddelenie, Žilina
- Spain (10):
  - Hospital Universitari de Bellvitge; Servicio de Oftalmologia, L'Hospitalet de Llobregat, Barcelona
  - Instituto Clinico Quirurgico de Oftalmologia - ICQO, Bilbao, Guipuzcoa
  - Instituto Oftalmologico Gomez Ulla, Santiago de Compostela, LA Coruña
  - Clinica Universitaria de Navarra; Servicio de Oftalmologia, Pamplona, Navarre
  - Hospital Perpetuo Socorro; Servicio de Oftalmología, Albacete
  - Institut de la Macula i la retina, Barcelona
  - Instituto de microcirugia ocular, Barcelona
  - VISSUM Madrid Santa Hortensia, Madrid
  - FISABIO. Fundación Oftalmologica del Mediterraneo, Valencia
  - Hospital Universitario Rio Hortega; Servicio de Oftalmologia, Valladolid
- Switzerland (3):
  - Inselspital Bern, Universitätsklinik für Augenheilkunde, Bern
  - Vista Klinik Binningen, Binningen
  - Stadtspital Triemli; Augenklinik, Zurich
- Turkey (Türkiye) (2):
  - Hacettepe University Medical Faculty, Ankara
  - Baskent University Ankara Hospital, Ankara
- United Kingdom (11):
  - Royal Victoria Hospital, Belfast
  - Bradford Royal Infirmary, Bradford
  - Bristol Eye Hospital, Bristol
  - University Hospital of Wales, Cardiff
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - Royal Liverpool University Hospital; St Paul's Clinical Eye Research Centre, Liverpool
  - Macular Treatment Centre; Royal Eye Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Southampton General Hospital, Southampton
  - The Royal Wolverhampton Hospitals NHS Trust, Wolverhampton
  - The York Hospital, York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 994 participants enrolled in study . study terminated early by Sponsor due to lack of efficacy.
  842 patients received at least one lampalizumab injection 152 patients enrolled in Study GX30191 did not receive study drug in the extension study and thus were excluded from the safety-evaluable population.
Pre-assignment Details: Eligible participants were those who enrolled in Studies GX29176 (NCT02247479) and GX29185 (NCT02247531) and had completed the 96-week treatment period without early treatment discontinuation or study discontinuation.
Groups:
- Lampalizumab Q4W - Treatment-Naive: Participants who received sham comparator every 4 weeks in one of the parent studies and completed the Week 96 visit received lampalizumab, 10 milligrams (mg), by intravitreal (ITV) injection, administered every 4 weeks.
- Lampalizumab Q4W - Previously Treated: Participants who received lampalizumab every 4 weeks in one of the parent studies and completed the Week 96 visit received lampalizumab, 10 mg, by ITV injection, administered every 4 weeks.
- Lampalizumab Q6W - Treatment-Naive: Participants who received sham comparator every 6 weeks in one of the parent studies and completed the Week 96 visit received lampalizumab, 10 mg, by ITV injection, administered every 6 weeks.
- Lampalizumab Q6W - Previously Treated: Participants who received lampalizumab every 6 weeks in one of the parent studies and completed the Week 96 visit received lampalizumab, 10 mg, by ITV injection, administered every 6 weeks.
Period: Overall Study
Arm/Group | Lampalizumab Q4W - Treatment-Naive | Lampalizumab Q4W - Previously Treated | Lampalizumab Q6W - Treatment-Naive | Lampalizumab Q6W - Previously Treated
Started | 145 | 274 | 146 | 277
Completed | 0 | 0 | 0 | 0
Not Completed | 145 | 274 | 146 | 277
Not completed — Adverse Event | 1 | 0 | 1 | 3
Not completed — Death | 3 | 3 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 15 | 8 | 14
Not completed — Study Terminated by Sponsor | 134 | 252 | 135 | 251
Not completed — Physician Decision | 0 | 2 | 2 | 2
Not completed — Reason Not Specified | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety-evaluable population included all participants who enrolled in the extension study and received at least one lampalizumab injection in the extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lampalizumab Q4W - Treatment-Naive | Lampalizumab Q4W - Previously Treated | Lampalizumab Q6W - Treatment-Naive | Lampalizumab Q6W - Previously Treated | Total
Number analyzed (Participants) | 145 | 274 | 146 | 277 | 842
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.0 (8.2) | 78.7 (7.8) | 79.2 (8.6) | 80.2 (7.9) | 79.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 167 | 79 | 164 | 492
  Male | 63 | 107 | 67 | 113 | 350
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 145 | 269 | 141 | 272 | 827
  Multiple | 0 | 0 | 2 | 2 | 4
  Unknown | 0 | 3 | 1 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 4 | 12 | 21
  Not Hispanic or Latino | 140 | 267 | 140 | 263 | 810
  Unknown | 3 | 2 | 1 | 1 | 7
  Not Reported | 0 | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ocular Adverse Events (AEs) by Severity
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, or any deterioration in a laboratory value or other clinical test. Ocular AEs are the events which are localized in the ocular region.
Time Frame: Up to approximately one year
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- All Participants: All participants in the study received lampalizumab 10 mg, ITV, Q4W or Q6W.
Arm/Group | Lampalizumab Q4W - Treatment-Naive | Lampalizumab Q4W - Previously Treated | Lampalizumab Q6W - Treatment-Naive | Lampalizumab Q6W - Previously Treated | All Participants
Number analyzed (Participants) | 145 | 274 | 146 | 277 | 842
percentage of participants
  Any severity | 37.2 | 40.1 | 24.7 | 33.2 | 34.7
  Mild | 25.5 | 26.6 | 16.4 | 21.7 | 23.0
  Moderate | 9.7 | 11.3 | 8.2 | 10.1 | 10.1
  Severe | 2.1 | 2.2 | 0 | 1.4 | 1.5

2. Primary Outcome: Percentage of Participants With Systemic (Non-Ocular) AEs by Severity
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, or any deterioration in a laboratory value or other clinical test.
Time Frame: Up to approximately one year
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Lampalizumab Q4W - Treatment-Naive | Lampalizumab Q4W - Previously Treated | Lampalizumab Q6W - Treatment-Naive | Lampalizumab Q6W - Previously Treated | All Participants
Number analyzed (Participants) | 145 | 274 | 146 | 277 | 842
percentage of participants
  Any severity | 55.2 | 54.0 | 41.8 | 51.3 | 51.2
  Mild | 18.6 | 20.1 | 17.8 | 20.9 | 19.7
  Moderate | 28.3 | 20.4 | 18.5 | 20.2 | 21.4
  Severe | 8.3 | 13.5 | 5.5 | 10.1 | 10.1

3. Primary Outcome: Percentage of Participants With Anti-Lampalizumab Antibodies
Description: The immunogenicity analysis included participants with at least one predose and one postdose anti-lampalizumab antibodies assessment. Predose was defined as prior to the first dose in the extension study for the prior sham participants, and prior to the first dose in the parent study for the prior lampalizumab participants.
Time Frame: Week 48
Population: The safety-evaluable population included all participants who enrolled in the extension study and received at least one lampalizumab injection in the extension study. Data is reported for evaluable participants.
Measure: Number; unit: percentage of participants
Arm/Group | Lampalizumab Q4W - Treatment-Naive | Lampalizumab Q4W - Previously Treated | Lampalizumab Q6W - Treatment-Naive | Lampalizumab Q6W - Previously Treated | All Participants
Number analyzed (Participants) | 145 | 274 | 146 | 277 | 842
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to approximately one year
Description: The safety-evaluable population included all participants who enrolled in the extension study and received at least one lampalizumab injection in the extension study.
Arm/Group | Lampalizumab Q4W - Treatment-Naive | Lampalizumab Q4W - Previously Treated | Lampalizumab Q6W - Treatment-Naive | Lampalizumab Q6W - Previously Treated | All Participants
All-Cause Mortality (participants affected / at risk) | 3/145 | 3/274 | 0/146 | 9/277 | 15/842
Serious Adverse Events (participants affected / at risk) | 31/145 | 58/274 | 14/146 | 50/277 | 153/842
Other Adverse Events (participants affected / at risk) | 41/145 | 63/274 | 26/146 | 56/277 | 186/842
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lampalizumab Q4W - Treatment-Naive (N=145) | Lampalizumab Q4W - Previously Treated (N=274) | Lampalizumab Q6W - Treatment-Naive (N=146) | Lampalizumab Q6W - Previously Treated (N=277) | All Participants (N=842)
Visual acuity reduced (Eye disorders) | 1 | 4 | 1 | 2 | 8
Neovascular age-related macular degeneration (Eye disorders) | 1 | 1 | 1 | 2 | 5
Ocular hypertension (Eye disorders) | 0 | 2 | 0 | 0 | 2
Visual impairment (Eye disorders) | 1 | 1 | 0 | 0 | 2
Dellen (Eye disorders) | 0 | 1 | 0 | 0 | 1
Dry age-related macular degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 1
Iritis (Eye disorders) | 0 | 1 | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 2
Intraocular pressure increased (Investigations) | 3 | 4 | 1 | 5 | 13
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3 | 0 | 1 | 6
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 4 | 4
Bradycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 3
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Malabsorption (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 2 | 1 | 1 | 5
Death (General disorders) | 1 | 0 | 0 | 3 | 4
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1
Sudden cardiac death (General disorders) | 0 | 1 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 2 | 2 | 5 | 12
Influenza (Infections and infestations) | 2 | 1 | 0 | 2 | 5
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 1 | 3
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Central nervous system infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Enterocolitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 4 | 1 | 5 | 10
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 1 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0 | 0 | 2
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dementia with lewy bodies (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Wernicke's encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 2
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Aortic calcification (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lampalizumab Q4W - Treatment-Naive (N=145) | Lampalizumab Q4W - Previously Treated (N=274) | Lampalizumab Q6W - Treatment-Naive (N=146) | Lampalizumab Q6W - Previously Treated (N=277) | All Participants (N=842)
Conjunctival haemorrhage (Eye disorders) | 17 | 17 | 12 | 20 | 66
Eye pain (Eye disorders) | 8 | 8 | 5 | 11 | 32
Nasopharyngitis (Infections and infestations) | 11 | 12 | 3 | 6 | 32
Fall (Injury, poisoning and procedural complications) | 11 | 12 | 5 | 14 | 42
Intraocular pressure increased (Investigations) | 2 | 23 | 5 | 17 | 47

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor because the compound had demonstrated lack of efficacy. Thus, no participant in this study completed the full duration of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT02745119/Prot_SAP_000.pdf